CLINICAL TRIAL: NCT01932450
Title: A Randomized, Open-label Study Investigating the Effect of Bilateral Renal Artery Sympathetic Denervation by Catheter-based Radiofrequency Ablation on Blood Pressure and Disease Progression in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Radiofrequency Ablation for ADPKD Blood Pressure and Disease Progression Control
Acronym: RAFALE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mei changlin (Other)
Responsible Party: Sponsor-Investigator, Mei changlin, Chief Physician, Professor, The director of Nephrology department and Internal Medicine department, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZKIPLA-ADPKD-001
Record Dates: First submitted 2013-08-18; First posted 2013-08-30 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Hypertension
Keywords: hypertension; radiofrequency ablation; autosomal dominant polycystic kidney disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic denervation (Experimental): One-time standard bilateral renal sympathetic denervation by catheter-based radiofrequency ablation and using antihypertensive drugs which at least include an angiotensin converting enzyme inhibitor (ACE-I) or an angiotensin II receptor blocker (ARB).
  Interventions: Procedure: renal sympathetic denervation; Drug: antihypertensive drugs
- antihypertensive drugs (Active Comparator): Blood pressure control in ADPKD patients with hypertension only using antihypertensive drugs which at least include an angiotensin converting enzyme inhibitor (ACE-I) or an angiotensin II receptor blocker (ARB)
  Interventions: Drug: antihypertensive drugs

INTERVENTIONS:
Procedure: renal sympathetic denervation — One-time standard Catheter-based renal sympathetic denervation will be performed in both renal arteries by radiofrequency ablation.
  Other Names: Percutaneous radiofrequency ablation of renal nerves; Transcatheter renal denervation; renal denervation; renal ablation
  Arms: renal sympathetic denervation
Drug: antihypertensive drugs — antihypertensive drugs have been used from baseline in patients, and will be modified by patient's blood pressure.

SUMMARY:
A randomized, open-label single-center study investigates the efficacy and safety of bilateral renal artery sympathetic denervation by catheter-based radiofrequency ablation on blood pressure and disease progression control in autosomal dominant polycystic kidney disease(ADPKD). The total number of study subjects will be 100. All of them have diagnosed with ADPKD and hypertension. Patients will be randomized 1:1 (50 with radiofrequency ablation(RFA), 50 only with drugs). Change in average office-based measurements of systolic blood pressure(SBP), average 24-hour systolic blood pressure by ambulatory blood pressure monitoring (ABPM) , incidence of office systolic blood pressure reductions of ≥10, ≥15 and ≥20 mm Hg , office diastolic blood pressure (DBP), number and dosage of blood pressure tablets, total kidney volume (TKV), total cyst volume (TCV), pain related to cystic kidneys and renal function, will be assessed at 12 months of follow-up. The safety variables will be assessed at every visit of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADPKD.
* Having hypertension, defined as systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg, and currently using 2 antihypertensive drugs and receiving a stable antihypertensive treatment regimen without change in dose or medication in the previous 30 days.
* Male and female patients 20 years to 60 years of age.
* Glomerular Filtration Rate (GFR) ≥30 ml/min/1.73 m2, estimated from serum creatinine using the Chronic Kidney Disease Epidemiology collaboration(CKD-EPI) equation.
* Have followed-up kidney and cyst volume at least 6 months in Shanghai Changzheng Hospital.
* Signed Informed Consent after being informed.

Exclusion Criteria:

* Documented renal vascular disease.
* Congenital absence of a kidney.
* Systemic illness with renal involvement.
* Spot urine albumin-to-creatinine ratio of >0.5 g/g and/or findings suggestive of kidney disease other than ADPKD.
* Exclusions specific to MRI acquisition and measurement: cardiac pacemaker, presence of MRI incompatible metallic clips or other material, excessive body weight, untreatable claustrophobia.
* Contraindications to the catheter-based renal denervation procedure by RFA, including allergy to radioiodinated contrast agents. Anatomical abnormalities of the renal arteries which preclude RFA: presence in either kidneys of multiple main renal arteries, main renal artery stenosis >50%, or main renal arteries of <4 mm in diameter or <20 mm in length.
* Contraindications on ethical grounds.
* Women who are pregnant or breast feeding.
* Intention to become pregnant during the course of the study.
* Lack of safe contraception: Female subjects of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Female subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential).
* Other clinically significant concomitant disease states (hepatic dysfunction, cardiovascular disease, metastatic cancer).
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
office-based measurements of systolic blood pressure | baseline and 12 months (day 360±14)
  Between-group change in average office-based measurements of systolic blood pressure from baseline to 12 months after randomization and One-time standard bilateral renal sympathetic denervation by catheter-based radiofrequency ablation.

SECONDARY OUTCOMES:
24-hour systolic blood pressure by ambulatory blood pressure monitoring (ABPM) | baseline and 12 months (day 360±14)
  Change in average 24-hour systolic blood pressure by ambulatory blood pressure monitoring (ABPM) from baseline to 12 month.
Incidence of office systolic blood pressure reduction | baseline and 12 months (day 360±14)
  Incidence of office systolic blood pressure reductions of ≥10, ≥15 and ≥20 mm Hg from baseline to 12 month.
office diastolic blood pressure | baseline and 12 months (day 360±14)
  Change in office diastolic blood pressure from baseline to 12 months.
number and dosage of blood pressure tablets | baseline and 12 months (day 360±14)
  Change in number and dosage of blood pressure tablets from baseline to 12 months.
estimated Glomerular Filtration Rate(eGFR) | baseline and 12 months (day 360±14)
  Change in estimated Glomerular Filtration Rate(eGFR) from baseline to 12 months.
albuminuria | baseline and 12 months (day 360±14)
  Change in albuminuria from baseline to 12 months.
total kidney volume (TKV) | baseline and 12 months (day 360±14)
  Change in total kidney volume (TKV) from baseline to 12 months
pain | baseline and 12 months (day 360±14)
  Change in pain related to cystic kidneys from baseline to 12 months.
procedure-related complications at femoral puncture site | up to 1 year (after radiofrequency ablation)
  Occurrence of procedure-related complications at femoral puncture site (hematoma, arteriovenous fistula, pseudoaneurysma).
Renal artery lesion | up to 1 year (after radiofrequency ablation)
  Renal artery lesion (perforation or dissection).
New renal artery stenosis | up to 1 year (after radiofrequency ablation)
  New renal artery stenosis >70%, determined by MRI within 12 months of randomization.
Embolic events | up to 1 year (after radiofrequency ablation)
  Embolic events.
hypotension | up to 1 year (after radiofrequency ablation)
  Episodes of hypotension.
hypertension. | up to 1 year (after radiofrequency ablation)
  Episodes of hypertension.
acute kidney injury | up to 1 year (after radiofrequency ablation)
  Acute deterioration of renal function
total cyst volume (TCV) | baseline and 12 months (day 360±14)
  Change in total cyst volume (TCV) from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, MD, Principal Investigator — Nephrology Department of Shanghai Changzheng Hospital
Locations (1):
- Department of Nephrology, Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Torres VE, Harris PC, Pirson Y. Autosomal dominant polycystic kidney disease. Lancet. 2007 Apr 14;369(9569):1287-1301. doi: 10.1016/S0140-6736(07)60601-1. PMID 17434405
- [Background] Harris PC, Torres VE. Polycystic kidney disease. Annu Rev Med. 2009;60:321-37. doi: 10.1146/annurev.med.60.101707.125712. PMID 18947299
- [Background] Grantham JJ. Clinical practice. Autosomal dominant polycystic kidney disease. N Engl J Med. 2008 Oct 2;359(14):1477-85. doi: 10.1056/NEJMcp0804458. No abstract available. PMID 18832246
- [Background] Chang MY, Ong AC. Autosomal dominant polycystic kidney disease: recent advances in pathogenesis and treatment. Nephron Physiol. 2008;108(1):p1-7. doi: 10.1159/000112495. Epub 2007 Dec 13. PMID 18075279
- [Background] Neumann J, Ligtenberg G, Klein IH, Blankestijn PJ. Pathogenesis and treatment of hypertension in polycystic kidney disease. Curr Opin Nephrol Hypertens. 2002 Sep;11(5):517-21. doi: 10.1097/00041552-200209000-00007. PMID 12187316
- [Background] Chapman AB, Johnson AM, Rainguet S, Hossack K, Gabow P, Schrier RW. Left ventricular hypertrophy in autosomal dominant polycystic kidney disease. J Am Soc Nephrol. 1997 Aug;8(8):1292-7. doi: 10.1681/ASN.V881292. PMID 9259356
- [Background] Ecder T, Schrier RW. Hypertension in autosomal-dominant polycystic kidney disease: early occurrence and unique aspects. J Am Soc Nephrol. 2001 Jan;12(1):194-200. doi: 10.1681/ASN.V121194. No abstract available. PMID 11134267
- [Background] Chapman AB, Stepniakowski K, Rahbari-Oskoui F. Hypertension in autosomal dominant polycystic kidney disease. Adv Chronic Kidney Dis. 2010 Mar;17(2):153-63. doi: 10.1053/j.ackd.2010.01.001. PMID 20219618
- [Background] Cerasola G, Vecchi M, Mule G, Cottone S, Mangano MT, Andronico G, Contorno A, Parrino I, Renda F, Pavone G. Sympathetic activity and blood pressure pattern in autosomal dominant polycystic kidney disease hypertensives. Am J Nephrol. 1998;18(5):391-8. doi: 10.1159/000013382. PMID 9730562
- [Background] Klein IHHT, Ligtenberg G, Oey PL, Koomans HA, Blankestijn PJ. Sympathetic activity is increased in polycystic kidney disease and is associated with hypertension. J Am Soc Nephrol. 2001 Nov;12(11):2427-2433. doi: 10.1681/ASN.V12112427. PMID 11675419
- [Background] Schrier RW. Hypertension and autosomal dominant polycystic kidney disease. Am J Kidney Dis. 2011 Jun;57(6):811-3. doi: 10.1053/j.ajkd.2011.02.379. No abstract available. PMID 21601126
- [Background] Chapman AB, Torres VE, Perrone RD, Steinman TI, Bae KT, Miller JP, Miskulin DC, Rahbari Oskoui F, Masoumi A, Hogan MC, Winklhofer FT, Braun W, Thompson PA, Meyers CM, Kelleher C, Schrier RW. The HALT polycystic kidney disease trials: design and implementation. Clin J Am Soc Nephrol. 2010 Jan;5(1):102-9. doi: 10.2215/CJN.04310709. PMID 20089507
- [Background] Torres VE, Chapman AB, Perrone RD, Bae KT, Abebe KZ, Bost JE, Miskulin DC, Steinman TI, Braun WE, Winklhofer FT, Hogan MC, Oskoui FR, Kelleher C, Masoumi A, Glockner J, Halin NJ, Martin DR, Remer E, Patel N, Pedrosa I, Wetzel LH, Thompson PA, Miller JP, Meyers CM, Schrier RW; HALT PKD Study Group. Analysis of baseline parameters in the HALT polycystic kidney disease trials. Kidney Int. 2012 Mar;81(6):577-85. doi: 10.1038/ki.2011.411. Epub 2011 Dec 28. PMID 22205355
- [Background] Gattone VH 2nd, Siqueira TM Jr, Powell CR, Trambaugh CM, Lingeman JE, Shalhav AL. Contribution of renal innervation to hypertension in rat autosomal dominant polycystic kidney disease. Exp Biol Med (Maywood). 2008 Aug;233(8):952-7. doi: 10.3181/0802-RM-54. Epub 2008 May 14. PMID 18480417
- [Background] Chapuis O, Sockeel P, Pallas G, Pons F, Jancovici R. Thoracoscopic renal denervation for intractable autosomal dominant polycystic kidney disease-related pain. Am J Kidney Dis. 2004 Jan;43(1):161-3. doi: 10.1053/j.ajkd.2003.07.026. PMID 14712440
- [Background] Valente JF, Dreyer DR, Breda MA, Bennett WM. Laparoscopic renal denervation for intractable ADPKD-related pain. Nephrol Dial Transplant. 2001 Jan;16(1):160. doi: 10.1093/ndt/16.1.160. No abstract available. PMID 11209012
- [Background] Hogan MC, Norby SM. Evaluation and management of pain in autosomal dominant polycystic kidney disease. Adv Chronic Kidney Dis. 2010 May;17(3):e1-e16. doi: 10.1053/j.ackd.2010.01.005. PMID 20439087
- [Background] MORRISSEY DM, BROOKES VS, COOKE WT. Sympathectomy in the treatment of hypertension; review of 122 cases. Lancet. 1953 Feb 28;1(6757):403-8. doi: 10.1016/s0140-6736(53)91589-x. No abstract available. PMID 13024041
- [Background] SMITHWICK RH, THOMPSON JE. Splanchnicectomy for essential hypertension; results in 1,266 cases. J Am Med Assoc. 1953 Aug 15;152(16):1501-4. doi: 10.1001/jama.1953.03690160001001. No abstract available. PMID 13061307
- [Background] EVELYN KA, SINGH MM, CHAPMAN WP, PERERA GA, THALER H. Effect of thoracolumbar sympathectomy on the clinical course of primary (essential) hypertension. A ten-year study of 100 sympathectomized patients compared with individually matched, symptomatically treated control subjects. Am J Med. 1960 Feb;28:188-221. doi: 10.1016/0002-9343(60)90184-4. No abstract available. PMID 13821037
- [Background] Schlaich MP, Sobotka PA, Krum H, Lambert E, Esler MD. Renal sympathetic-nerve ablation for uncontrolled hypertension. N Engl J Med. 2009 Aug 27;361(9):932-4. doi: 10.1056/NEJMc0904179. No abstract available. PMID 19710497
- [Background] Schlaich MP, Hering D, Sobotka P, Krum H, Lambert GW, Lambert E, Esler MD. Effects of renal denervation on sympathetic activation, blood pressure, and glucose metabolism in patients with resistant hypertension. Front Physiol. 2012 Feb 2;3:10. doi: 10.3389/fphys.2012.00010. eCollection 2012. PMID 22347190
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Symplicity HTN-1 Investigators. Catheter-based renal sympathetic denervation for resistant hypertension: durability of blood pressure reduction out to 24 months. Hypertension. 2011 May;57(5):911-7. doi: 10.1161/HYPERTENSIONAHA.110.163014. Epub 2011 Mar 14. PMID 21403086
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Background] Kandzari DE, Bhatt DL, Sobotka PA, O'Neill WW, Esler M, Flack JM, Katzen BT, Leon MB, Massaro JM, Negoita M, Oparil S, Rocha-Singh K, Straley C, Townsend RR, Bakris G. Catheter-based renal denervation for resistant hypertension: rationale and design of the SYMPLICITY HTN-3 Trial. Clin Cardiol. 2012 Sep;35(9):528-35. doi: 10.1002/clc.22008. Epub 2012 May 9. PMID 22573363
- [Background] Hering D, Mahfoud F, Walton AS, Krum H, Lambert GW, Lambert EA, Sobotka PA, Bohm M, Cremers B, Esler MD, Schlaich MP. Renal denervation in moderate to severe CKD. J Am Soc Nephrol. 2012 Jul;23(7):1250-7. doi: 10.1681/ASN.2011111062. Epub 2012 May 17. PMID 22595301
- [Background] Casale P, Meyers K, Kaplan B. Follow-up for laparoscopic renal denervation and nephropexy for autosomal dominant polycystic kidney disease-related pain in pediatrics. J Endourol. 2008 May;22(5):991-3. doi: 10.1089/end.2007.0359. PMID 18370613
- [Background] Schlaich MP, Krum H, Esler MD. New therapeutic approaches to resistant hypertension. Curr Hypertens Rep. 2010 Aug;12(4):296-302. doi: 10.1007/s11906-010-0119-1. PMID 20509010
- [Background] Serra AL, Poster D, Kistler AD, Krauer F, Raina S, Young J, Rentsch KM, Spanaus KS, Senn O, Kristanto P, Scheffel H, Weishaupt D, Wuthrich RP. Sirolimus and kidney growth in autosomal dominant polycystic kidney disease. N Engl J Med. 2010 Aug 26;363(9):820-9. doi: 10.1056/NEJMoa0907419. Epub 2010 Jun 26. PMID 20581391
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Celermajer DS. Testing endothelial function using ultrasound. J Cardiovasc Pharmacol. 1998;32 Suppl 3:S29-32. PMID 9883744
- [Background] Deanfield J, Donald A, Ferri C, Giannattasio C, Halcox J, Halligan S, Lerman A, Mancia G, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Schiffrin EL, Taddei S, Webb DJ; Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part I: Methodological issues for assessment in the different vascular beds: a statement by the Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Jan;23(1):7-17. doi: 10.1097/00004872-200501000-00004. PMID 15643116
- [Background] Gemignani V, Bianchini E, Faita F, Giannarelli C, Plantinga Y, Ghiadoni L, Demi M. Ultrasound measurement of the brachial artery flow-mediated dilation without ECG gating. Ultrasound Med Biol. 2008 Mar;34(3):385-91. doi: 10.1016/j.ultrasmedbio.2007.08.006. Epub 2007 Oct 26. PMID 17964069
- [Background] Sudano I, Flammer AJ, Periat D, Enseleit F, Hermann M, Wolfrum M, Hirt A, Kaiser P, Hurlimann D, Neidhart M, Gay S, Holzmeister J, Nussberger J, Mocharla P, Landmesser U, Haile SR, Corti R, Vanhoutte PM, Luscher TF, Noll G, Ruschitzka F. Acetaminophen increases blood pressure in patients with coronary artery disease. Circulation. 2010 Nov 2;122(18):1789-96. doi: 10.1161/CIRCULATIONAHA.110.956490. Epub 2010 Oct 18. PMID 20956208
- [Background] Williams B, Lacy PS, Thom SM, Cruickshank K, Stanton A, Collier D, Hughes AD, Thurston H, O'Rourke M; CAFE Investigators; Anglo-Scandinavian Cardiac Outcomes Trial Investigators; CAFE Steering Committee and Writing Committee. Differential impact of blood pressure-lowering drugs on central aortic pressure and clinical outcomes: principal results of the Conduit Artery Function Evaluation (CAFE) study. Circulation. 2006 Mar 7;113(9):1213-25. doi: 10.1161/CIRCULATIONAHA.105.595496. Epub 2006 Feb 13. PMID 16476843
- [Background] Pannier B, Guerin A, London G, Asmar R, Safar M; REASON Study. [Combination of low-dose perindopril/indapamide versus atenolol in the hypertensive patient. Effects on systolic pressure and arterial hemodynamics. REASON Study]. Arch Mal Coeur Vaiss. 2002 Sep;95 Spec No 6:11-6. French. PMID 12407781
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039